CLINICAL TRIAL: NCT06212557
Title: Evaluation of KIOS in a 12-week Randomized Controlled Trial
Brief Title: KIOS Mobile App Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Biomedical Development Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20210407H; R42DA054881 (NIH)
Record Dates: First submitted 2024-01-08; First posted 2024-01-19 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder
Keywords: Digital health therapeutic; Behavioral intervention strategies; Clinic-based counseling
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled 2 arm trial
Who Masked: Investigator
Masking Description: Randomization will be stratified by two characteristics: (1) history of MOUD and (2) stimulant use in past one month. Allocation to treatment groups will be randomly assigned by 1:1 allotment to either KIOS + TAU (treatment as usual) or KIOS sham + TAU with strata. Study staff will be blind to the condition to which the participant is assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Treatment as Usual plus KIOS App (Experimental): Treatment as usual in clinics with the use of the KIOS App
  Interventions: Device: KIOS App; Behavioral: Treatment as usual
- Treatment as Usual plus KIOS education App (Sham Comparator): Treatment as usual in clinics with the use of the KIOs education App (Sham)
  Interventions: Behavioral: KIOS App education; Behavioral: Treatment as usual

INTERVENTIONS:
Device: KIOS App — KIOS provides patients on demand individualized advice and reinforcement of lifestyle interventions to improve self-management during Medication-Assisted Treatment (MAT)
  Other Names: KIOS
  Arms: Active Treatment as Usual plus KIOS App
Behavioral: KIOS App education — Educational tools provided to participants with opioid use disorder
  Other Names: KIOS education
  Arms: Treatment as Usual plus KIOS education App
Behavioral: Treatment as usual — Behavioral counseling in clinic
  Other Names: TAU

SUMMARY:
Evaluation of a mobile medical app (KIOS) vs. treatment as usual for the treatment of opioid use disorder (OUD).

DETAILED DESCRIPTION:
The study is a parallel intervention examining the KIOS app, a digital health therapeutic intended to help individuals in recovery from opioid use disorder better self-manage their condition. KIOS will offer individualized, evidence-based behavioral intervention strategies responsive to the patients' current clinical status outside the setting of the doctor's office or treatment facility. KIOS makes it possible to process patient-entered data and provide responsive behavioral advice to patients specific to their condition in real time. KIOS gives patients 24/7 access to behavioral intervention strategies that can augment and improve response to routine clinic-based counseling interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients 18 years of age or older
2. Patients must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
3. DSM-5 (Diagnostic and Statistical Manual of Mental Disorders fifth edition) criteria for opioid use disorder
4. Ability to access KIOS via smartphone or tablet
5. Recently (less than 6 months) enrolled in and currently participating in MOUD at a clinic in Texas

Exclusion Criteria:

1. Unwilling or unable to comply with study requirements
2. Psychiatric or medical disorder interfering with ability to use the app
3. Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Retention in treatment | Baseline to 13 weeks
  Measured by the number of days from the start of the 13-week intervention until the participant either leaves the trial, or completes the trial

SECONDARY OUTCOMES:
Measure of opioid use reduction | 60 days to 13 weeks
  Defined as abstaining from opioids during the last week and for at least 2 of the previous 3 weeks of the third month of MOUD treatment
Percentage of Opioid Abstinent Days | Baseline to 13 weeks
  Total abstinence, measured by urinalysis confirmed self-report of opioid use during the 13-week intervention
Completion of treatment | Baseline to 13 weeks
  Number of subjects that completed their participation in the study
Patient Health Questionnaire-9 (PHQ-9) | Baseline and 13 weeks
  A 9 item questionnaire scored from 0 (Not at all) to 4 (Nearly every day) with a potential score of 0-36 with a lower score indicating better health and emotional well-being.
Treatment Effectiveness Assessment TEA) | Baseline and 13 weeks
  The TEA asks the participant to express the extent of changes for the better from your involvement in the program to this point (or how things are if it's your first TEA or baseline) in four areas: substance use, health, lifestyle, and community. For each area, think about how things have become better and circle the results on the scale below: the more you have improved, the higher the number -from 1 (not better at all) to 10 (very much better). Possible scores are between 1 and 40 with a lower score indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Potter, PhD, MPH, Principal Investigator — The University of Texas Health Science Center at San Antonio; Elise Marino, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center - Department of Psychiatry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will be conducted in accordance with the following publication and data sharing policies and regulations:
  National Institutes of Health (NIH) Public Access Policy, which ensures that the public has access to the published results of NIH funded research. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive PubMed Central upon acceptance for publication.
  This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study completion and data analysis when summary results are posted on ClinicalTrials.gov and then after peer review and publication acceptance.